CLINICAL TRIAL: NCT02073071
Title: Effects of Infant Formula on the Growth and Tolerance in Preterm/Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA05
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Other Preterm Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm/low birth weight infants: Preterm infant formula per standard of care
  Interventions: Other: Preterm infant formula per standard of care

INTERVENTIONS:
Other: Preterm infant formula per standard of care — Commercially available preterm infant formula

SUMMARY:
This is a two stage open-label, single-arm, multicenter and observational study.

DETAILED DESCRIPTION:
Stage 1: In hospital, preterm/low birth weight infants less than or equal to 34 weeks gestational age at birth, birth weight of ≥ 1000g to <1800g and conditions meeting the enrollment criteria will be fed formula with or without parenteral nutrition until discharge. Stage 2: Post-discharge, all infants with birth weight < or =1500g will be followed on formula per standard of care and accepted standard of care including feeding until the infant's weight >or= 25th percentile of growth expectation based on corrected age (P25) or until infant reaches 9 months corrected age.

ELIGIBILITY:
Inclusion Criteria for Stage 1:

* Less than or equal to 34 weeks gestational age at birth, and birth weight ≥ 1000g to < 1800g;
* Apgar score in 5 minutes after birth ≥ 7;
* Infant is 21 days or less of age at enrollment;
* Only singleton or twin births;
* Infants who can receive early enteral feeding stably (reaching 50% or higher of the required daily total calories) and whose parents/guardians and investigators have selected Similac Special Care (SSC) for feeding;
* Infant has been classified as appropriate for gestational age (AGA) or if classified as asymmetric small for gestational age (SGA) (Asymmetric SGA: Weight below the 10th percentile, but head circumference is greater than or equal to the 10th percentile) enrollment has been preapproved by sponsor;

Inclusion Criteria for Stage 2:

* Infants with birth weight < or = 1500g, subjects whose parents/guardians and investigators have selected NeoSure for continued feeding after hospital discharge.

Exclusion Criteria for Stage 1:

* Serious congenital chromosomal or metabolic abnormalities that may affect growth and development;
* Congenital gastrointestinal malformations , including but not limited to congenital megacolon or gastric-intestinal perforation;
* Serious complications associated with preterm birth, including but not limited to necrotizing enterocolitis (NEC), septicemia or sepsis;
* Other serious disorders of cardiac/respiratory/endocrine/hematological/ gastrointestinal/other systems, or serious diseases requiring surgical intervention;
* Maternal incapacity: including maternal drug, cocaine or alcohol abuse during pregnancy or current;
* Infants who received any experimental treatment, participated in other clinical trials or received other study interventions unrelated to this study within 30 days prior to enrollment;
* Infants who have received or planned to receive breastfeeding or other infant formula (powder) other than SSC with calories intake ≥25% of the required daily total calories
* Intubation for ventilation at the time of enrollment.

Exclusion Criteria for Stage 2:

* Infants who have received breastfeeding or other infant formula (powder) during hospitalization other than SSC with calories intake ≥25% of the required daily total calories
* Infants who have planned to receive breastfeeding or other infant formula (powder) other than NeoSure after discharge with calories intake ≥25% of the required daily total calories

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospital based preterm infants
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Weight | Change from first feeding to discharge (up to ~8 weeks)

SECONDARY OUTCOMES:
Length | Change from first feeding to discharge (up to ~8 weeks)
Head Circumference | Change from first feeding to discharge (up to ~8 weeks)
Hospitalization Length of Stay | Time from Birth to discharge (up to ~8 weeks)
Gastrointestinal Tolerance | From first feeding to discharge (up to ~8 weeks)
  vomiting, abdominal distension, gastric residuals, stool abnormalities, necrotizing enterocolitis
Catch Up Growth | From discharge to 9 months corrected age
  From discharge to the time point that infant's weight >or= 25th percentile of growth expectation based on corrected age (P25) or until infant reaches 9 months corrected age.

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng Zhao, MD, PhD, Study Chair — Abbott Nutrition China
Locations (10):
- China (10):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hunan Children's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Children's hospital of Chongqing Medical University, Chongqing
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Center Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai